CLINICAL TRIAL: NCT01913756
Title: Dairy Products and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Life Sciences (Other)
Collaborators: Tine (Industry)
Responsible Party: Principal Investigator, Rita Nilsen, PhD Student, Norwegian University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REK-340857
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Blood Pressure; Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Gouda-type cheese (Experimental): 80 g/day Gouda-type cheese
  Interventions: Dietary Supplement: Gouda-type cheese
- Low cheese intake (No Intervention)
- Gamalost (Norwegian traditional cheese) (Experimental): 50 g/day Gamalost
  Interventions: Dietary Supplement: Gamalost (Norwegian traditional cheese)

INTERVENTIONS:
Dietary Supplement: Gamalost (Norwegian traditional cheese)
  Arms: Gamalost (Norwegian traditional cheese)
Dietary Supplement: Gouda-type cheese
  Arms: Gouda-type cheese

SUMMARY:
The purpose of this trial is to investigate the effect of dairy products on the so called metabolic syndrome. Metabolic syndrome is a cluster of risk factors, such as high blood pressure and high cholesterol, for the development of diabetes and heart disease. Participants will be randomly assigned to either eat a portion of a Norwegian traditional cheese which is high in protein and low in fat (group 1), or eat a slightly higher than normal intake of regular Gouda-type cheese (group 2), or to limit their intake of cheese (group 3).

Dairy products are a significant source of bioactive peptides, small pieces of protein which may have an effect on our health. These effects may be antimicrobial, antioxidative, or blood pressure lowering. The traditional Norwegian cheese, Gamalost, which is naturally high in protein (50%) and low in fat (<1%), has been found to be particularly high in these bioactive peptides. Specifically, the cheese was found to have a very high ACE-inhibitory activity, meaning it has the potential to lower blood pressure without the use of pharmaceuticals.

A pilot study was performed in May 2012. No intervention was given in this trial, but participants answered an extensive questionnaire about dietary habits and lifestyle. This trial found that the people who ate the most Gamalost had a slightly lower blood pressure than those that did not eat the cheese. Since that was just a point-in-time study with no intervention or control, the investigators are not able to say anything certain about cause and effect, which is why the investigators want to perform this larger controlled study.

In total, the investigators aim to recruit 300 people to participate in this trial, i.e. 100 in each group. The participants will be randomly placed in one of the groups and they will have to do the intervention for eight weeks. At inclusion, the investigators measure blood pressure, fasting blood glucose, weight, height, waist circumference, and the investigators draw a fasting blood sample to measure cholesterol. The same measurements will be repeated at the end of the eight weeks. At inclusion they will also fill out an extensive questionnaire about their diet and lifestyle. A shorter version of the same questionnaire will also be given at the end of the trial period.

The overall goal of the study is to assess the effect of dairy products on the metabolic syndrome, but the main hypothesis is to assess whether a high intake of Gamalost can reduce blood pressure in a group of people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Must be able to eat cheese evey day

Exclusion Criteria:

* Pregnant women
* Taking blood pressure lowering medication
* Not able to read Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline, 4 weeks and 8 weeks.

SECONDARY OUTCOMES:
Change in serum cholesterol levels | Baseline and 8 weeks.
Change in body composition. | Baseline and 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian University of Life Sciences, Aas, Aas, Norway